CLINICAL TRIAL: NCT02111317
Title: A Phase 1, Open-label, Single-Sequence, Crossover Drug Interaction Study to Evaluate the Effect of Verapamil on the Pharmacokinetics of ASP015K in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Verapamil on the Pharmacokinetics of ASP015K in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Janssen Biotech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 015K-CL-PK04
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Healthy Subjects; Pharmacokinetics of ASP015K
Keywords: ASP015K; Pharmacokinetics; Healthy Subjects
MeSH Terms: interventions — peficitinib; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP015K and verapamil (Experimental): Single dose of ASP015K, then repeat dose of verapamil, then a second single dose of ASP015K while continuing verapamil
  Interventions: Drug: ASP015K; Drug: verapamil

INTERVENTIONS:
Drug: ASP015K — oral
Drug: verapamil — oral
  Other Names: CALAN®

SUMMARY:
The purpose of this study is to evaluate the effect of verapamil, a P-glycoprotein (P-gp) inhibitor, on the pharmacokinetics of ASP015K. This study will also assess the safety and tolerability of ASP015K administered alone and also and in combination with verapamil.

DETAILED DESCRIPTION:
Eligible subjects will be admitted to the clinical unit on day -1 and remain confined until day 15.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a Body Mass Index (BMI) range of 18.5-32.0 kg/m2, inclusive, and must weigh at least 50 kg
* Subject must be capable of swallowing multiple tablets
* Subject agrees not to participate in another investigational study while on treatment

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to verapamil, ASP015K, or any components of the formulations used.
* Subject has any of the liver function tests above the upper limit of normal (ULN)
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Subject has any history or evidence of any clinically significant cardiovascular, GI, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, and/or other major disease or malignancy
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory) infection, or fungal (noncutaneous) infection within 1 week prior to day -1.
* Subject has any clinically significant abnormality following physical examination, ECG, such as sick sinus syndrome, second- or third-degree atrioventricular block, or atrial flutter/atrial fibrillation, or clinical laboratory tests
* Subject has a mean pulse < 50 or > 90 beats per minute (bpm); mean systolic blood pressure (SBP) < 100 or > 140 mmHg; mean diastolic blood pressure (DBP) < 60 or > 90 mmHg (measurements taken in triplicate after subject has been resting in sitting position for 5 minutes)
* Subject has a mean QTcF interval of > 430 msec (for males) and > 450 msec (for females)
* Subject has used any prescribed or nonprescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's Wort) in the 2 weeks prior to study drug administration, with the exception of hormone replacement therapy (HRT) and intermittent acetaminophen (no more than 2 g per day)
* Subject has smoked or has used tobacco-containing products and nicotine or nicotine-containing products in the past 6 months
* Subject has a history of consuming more than 14 units of alcoholic beverages per week within 6 months prior to screening or has a history of alcoholism or drug/chemical substance abuse within past 2 years prior to screening (Note: one unit = 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits)
* Subject has a positive test for alcohol, drugs of abuse, or cotinine
* Subject anticipates an inability to abstain from xanthine (e.g., caffeine), grapefruit, Seville oranges (including marmalade), star fruit, or any products containing these items from 72 hours prior to day -1 and throughout the duration of the study
* Subject has used any inducer of metabolism (e.g., barbiturates, rifampin) in the past 3 months prior to day -1
* Subject has had any significant blood loss, donated 1 unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within past 7 days
* Subject has a positive test for hepatitis B surface antigen (HBsAg), anti-hepatitis A virus (Immunoglobulin [Ig] M), anti-hepatitis C virus (HCV), hepatitis B core antibody or anti-human immunodeficiency virus (HIV) type 1 or type 2
* Subject has a positive tuberculosis (TB) skin test, Quantiferon Gold® test or T-SPOT® test
* Subject received any vaccine within 60 days prior to study drug administration
* Subject has an absolute neutrophil count (ANC) < 2000 cells/mm3 or a creatine phosphokinase (CPK) > 1.5 x ULN
* Subject has had major gastrointestinal (GI) surgery or has a medical condition, which may inhibit the absorption and/or metabolism of study drug
* Subject has participated in any interventional clinical study or has been treated with any investigational drugs within 30 days or 5 half-lives of the drug, whichever is longer

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of ASP015K: Maximum concentration (Cmax) | Days 1-4 and Days 12-15
Pharmacokinetics of ASP015K: Area under the concentration-time curve (AUC) from time of dosing to the last quantifiable concentration (AUClast) | Days 1-4 and Days 12-15
Pharmacokinetics of ASP015K: AUC from the time of dosing extrapolated to time infinity (AUCinf) | Days 1-4 and Days 12-15

SECONDARY OUTCOMES:
Pharmacokinetic profile of ASP015K: time of maximum plasma concentration (tmax), terminal elimination half-life (t½), apparent total systemic clearance (CL/F), and apparent volume of distribution during the terminal elimination phase (Vz/F) | Days 1-4 and Days 12-15
Pharmacokinetic profile of ASP015K metabolites: Cmax, AUClast, AUCinf, tmax and t½ | Days 1-4 and Days 12-15

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Pharmacology Lead, Study Chair — Astellas Pharma Global Development, Inc.
Locations (1):
- PAREXEL, Glendale, California, United States